CLINICAL TRIAL: NCT06973707
Title: Digital Tools to Engage and Activate Patients During Hospitalization: A Cluster Randomized Trial
Brief Title: Digital Tools to Engage and Activate Patients During Hospitalization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Research Director, Division of General Internal Medicine, Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025p000989; R21HS030738 (Other Grant/Funding Number: AHRQ)
Record Dates: First submitted 2025-04-29; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hospital Information Systems
Keywords: Hospitalization; Health information technologies; Patient Engagement; Patient Activation
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Access to hospital's patient portal. Written materials regarding patient portal and structure of inpatient medical service. White board with plan of the day.
- Passive Digital Tools Only (Active Comparator): Usual Care plus: Dynamic organizational chart of care team members. Electronic guide to general medicine service. Electronic Plan for the Day.
  Interventions: Behavioral: Passive Digital Tools
- Passive Plus Active Digital Tools (Experimental): Usual Care plus Passive Tools plus: guide to why patient engagement is important. Sample medical questions with customized answers. Ability to create, organize, and store questions to ask the medical team. Electronic journal to keep track of symptoms, emotions, function, what patient learned.
  Interventions: Behavioral: Passive Digital Tools; Behavioral: Active Digital Tools

INTERVENTIONS:
Behavioral: Passive Digital Tools — Dynamic organizational chart of care team members Guide to general medicine service Plan for the day
  Arms: Passive Digital Tools Only; Passive Plus Active Digital Tools
Behavioral: Active Digital Tools — Guide: why patient engagement is important Sample questions with answers Ability to create, organize, and store questions to ask the medical team; reminder to ask them during rounds Electronic journal function with categories: symptoms, emotions, function, what I learned; reminder to share with medical team during rounds
  Arms: Passive Plus Active Digital Tools

SUMMARY:
The goal of this clinical trial is to learn about the possible benefits of mobile digital tools used by patients and families, with the help of a digital navigator, while patients are in the hospital. The goals are to better engage patients and their caregivers in their own care. The main questions it aims to answer are:

Will use of these digital tools and digital navigators lead to greater patient activation during the hospitalization than usual care? Will use of passive and active tools lead to greater patient activation than the use of passive tools alone? Will use of these digital tools increase patient knowledge (of the care team and care plan) and patient self-efficacy, reduce patient anxiety, and improve patient experience and post-discharge behavior (filling discharge prescriptions and keeping follow-up appointment visits)? Will use of the digital tools decrease disparities in outcomes by language and area deprivation index?

Participants will:

Be asked to use the digital tools, assisted by a digital navigator, or usual care, including the hospital's patient portal.

Complete surveys while in the hospital regarding baseline characteristics and study outcomes.

If asked, give input into the design of tools and/or participate in interviews regarding their opinions of the digital tools and any barriers to implementation.

DETAILED DESCRIPTION:
Patient activation, defined as having the knowledge, skills, and confidence to manage one's health condition, allows patients to better manage their medical symptoms and conditions, engage in activities that benefit their health, be involved in shared decision-making, and navigate the health care system. In the hospital, patient activation is often low. As a result, patients may receive suboptimal care during and after hospitalization. Digital tools such as patient portals have shown some promise to increase patient activation, but few studies have been conducted in the inpatient setting or have shown equivocal results due to low digital literacy.

The broad, long-term objectives of this work are to develop patient-facing digital tools, and assist patients with using them, in the hospital setting to increase patient activation and improve quality of care. The specific aims are: 1) Design and develop two sets of digital tools, passive and active, to better engage patients and their caregivers while in the hospital; 2) Pilot implementation of the two digital interventions on general medicine; and 3) Evaluate the effect of passive and active digital tools and digital navigators on patient activation, knowledge, and self-efficacy, patient behavior, patient experience, and equity.

During the R21 phase of the study, digital tools, built on top of the existing patient portal, will be developed and iteratively refined using user-centered design principles, with extensive input from patients, caregivers, and providers. Passive tools will provide additional information not available in our current patient portal, such as a dynamic organizational chart of each patient's care team. Active tools will provide customized answers to commonly asked questions and encourage patients to participate in their care, e.g., to ask their own questions during rounds and to keep (and share) a journal of their symptoms, function, and mood. A digital navigator will be recruited and trained to assist patients with the tools. Feasibility, acceptability, appropriateness, and usability will be evaluated using mixed methods, and a final implementation plan will be created. During the subsequent R33 phase, outcomes will be evaluated in a three-arm cluster-randomized controlled trial: usual care, passive tools only, or passive and active tools. Outcomes will include patient activation, patient experience, and downstream behaviors such as filling discharge prescriptions and keeping follow-up appointments. Mixed methods will be used to evaluate the reliability, validity, and usability of the tools and their impact on clinicians. An implementation guide will be created to facilitate widespread adoption and sustainability based on an evaluation of barriers and facilitators of implementation. Study findings will be disseminated to a variety of stakeholders to further the impact of this project on future care delivery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the general medicine service at Brigham and Women's Hospital during the 12-month trial enrollment period
* English or Spanish speakers
* Age 18 or older
* Able to provide informed consent

Exclusion Criteria:

* Residence in a nursing home, rehab facility, or group home
* Undomiciled
* Pregnant women, prisoners, or institutionalized individuals
* Dementia
* Likely to be discharged somewhere other than home in the opinion of the care team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2028-07-01 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in patient activation | Hospitalization (up to 30 days)
  Analytic variable: Patient Activation Measure (PAM)-13 day prior to discharge minus PAM-13 at enrollment. PAM-13 ranges from 0 to 100, with higher scores indicating greater patient activation (better outcome).
  Data source/method: survey

SECONDARY OUTCOMES:
Knowledge of care team | Day prior to discharge
  Analytic variable: Patient's knowledge of who is in charge of their care (Yes/No) Data source/method: survey
Knowledge of care plan | Day prior to discharge
  Analytic variable: Patient's knowledge of the plan for their care (Yes/No) Data source/method: survey
Self-efficacy for managing chronic conditions | Day prior to discharge
  Analytic variable: PROMIS Self-efficacy for managing chronic conditions score. T-score of 50 is average, standard deviation 10, higher scores indicate higher self-efficacy.
  Data source/method: survey
Improvement in anxiety and depression | Hospitalization (up to 30 days)
  Analytic variable: Hospital Anxiety Depression Scale (HADS) day prior to discharge minus HADS at enrollment. HADS consists of 14 questions with two subscales with 7 questions each for anxiety and depression. Each item is rated 0-3, resulting in a total score of 0-21 for each subscale, with higher scores indicating greater anxiety and depression.
  Data source/method: survey
Patient experience | Day prior to discharge
  Analytic variable: Picker Patient Experience Questionnaire score. 15 questions, each scored 1-5, with higher scores indicating greater patient experience.
  Data source/method: survey

OTHER OUTCOMES:
Post-discharge medication adherence | 0-3 days after discharge
  Analytic variable: Proportion of new medication prescriptions at discharge filled in the 3 days after discharge Data source/method: EHR discharge data, SureScripts prescription fill data
Keeping post-discharge appointments | 0-30 days after discharge
  Analytic variable: Proportion of scheduled appointments kept in the 30 days after discharge Data source/method: EHR appointment data

IPD SHARING:
Plan to Share IPD: Yes
Patient-level demographic data (from the EHR and patient survey). Outcome data (e.g., quality, safety, patient experience, equity) from patient surveys.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study data will be made available as soon as possible and no later than one year after the end of the award period. Data will be available for 10 years.
Access Criteria: Data will be restricted using a controlled access repository. Requests for data will be reviewed by the Co-PIs per established policies and procedures; the investigators may establish data use restrictions (e.g., only for research studies); a data user's institution will need to complete a Data Use Agreement; data users may need to produce a data security plan.